CLINICAL TRIAL: NCT04332744
Title: A Randomized Phase II Trial to Evaluate the Antitumor Activity of Enzalutamide and Talazoparib (PF-06944076) for the Treatment of Metastatic Hormone-naïve Prostate Cancer
Brief Title: Enzalutamide Plus Talazoparib for the Treatment of Hormone Sensitive Prostate Cancer (ZZ-First)
Acronym: ZZ-First
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP234; 2019-003096-20 (EudraCT Number)
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Prostate Cancer
Keywords: Prostate cancer; Metastatic prostate cancer; Hormone naïve; Unresectable prostate cancer; mHNPC; Prostate cancer stage IV; Prostatic neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; talazoparib

STUDY DESIGN:
Intervention Model Description: Randomized 1:2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Arm A) (Active Comparator): Patients will receive enzalutamide capsules orally once daily continuously (160 mg) in addition to standard ADT (unless surgical castration).
  Interventions: Drug: Enzalutamide
- Interventional Arm (Arm B) (Experimental): Patients will receive enzalutamide capsules 160 mg in combination with talazoparib (PF-06944076) capsules 0.5 mg, both orally daily and continuously in 28-day cycle, in addition to standard ADT (unless surgical castration).
  Interventions: Drug: Enzalutamide; Drug: Talazoparib

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide capsules orally once daily and continuously (160 mg) in 28-day cycles (every four weeks)
  Other Names: Xtandi
Drug: Talazoparib — Talazoparib capsules orally once daily and continuously (0.5 mg) in 28-day cycles (every four weeks)
  Other Names: (PF-06944076)
  Arms: Interventional Arm (Arm B)

SUMMARY:
This is a multicenter, open-label, randomized, two-arm, phase II clinical trial to evaluate the efficacy and safety of talazoparib (PF-06944076) in combination with enzalutamide in patients with metastatic hormone-naïve prostate cancer (mHNPC)

DETAILED DESCRIPTION:
Men age ≥ 18 years with high-volume mHNPC that are not candidates for curative intent and have not received previous systemic treatment with any other agent for unresectable locally advanced or mHNPC.

After signing ICF and confirm eligibility, patients will start treatment with enzalutamide in addition to standard ADT. After 2 cycles of enzalutamide-containing regimen, patients will be randomized in a 1:2 ratio to:

Cohort A - Enzalutamide 160 mg orally daily continuously; Cohort B - Enzalutamide 160 mg in combination with talazoparib (PF-06944076) 0.5 mg, both orally daily and continuously in 28-day cycles.

In either arm, patients will be requested to continue ADT throughout trial participation (unless surgical castration).

Randomization will be stratified based on HR gene alterations (presence versus absence/unknown) detected in the baseline biopsy.

Patients will receive treatment until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

Patients discontinuing the study treatment period will enter a post-treatment follow-up period during which survival and at least the first two new anti-cancer therapies will be collected every six months (± 14 days) from the last dose of investigational product until the end of study (EoS).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 y.o.) who signed informed consent form (ICF) prior to participation in any study-related activities.
2. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. High-volume metastatic disease documented on bone scan or computed tomography (CT)/magnetic resonance imaging (MRI) scan, defined as the presence of either visceral disease and/or at least four bone metastases on bone scan, with at least one of them beyond spine/pelvis.
5. Life expectancy of ≥ 12 months.
6. Histologically confirmed adenocarcinoma of the prostate without predominance of small-cell or neuroendocrine features according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines based on local testing on the most recent analyzed biopsy.

   Note: Central confirmation of adenocarcinoma is not required for study entry. However, tissue blocks, or slides, must be submitted to confirm the diagnoses by a Sponsor-designated central laboratory retrospectively and/or exploratory biomarker analyses.
7. Willingness and ability to provide tumor paired biopsies during the study participation in order to perform exploratory studies. At the study entry, the most recent tumor biopsy since last progression from either metastatic or primary tissues will be provided. If not feasible, patient eligibility should be evaluated by a Sponsor's qualified designee.
8. Adequate hematologic and organ function within 28 days before the first study treatment on Cycle 1 Day 1, defined by the following:

   1. Hematological: White blood cell (WBC) count > 3.0 x 109/L; Absolute neutrophil count (ANC) > 1.5 x 109/L; Platelet count > 100.0 x109/L; Hemoglobin (Hb) > 9.0 g/dL.

      Note: Patients receiving growth factors or blood transfusions within 14 days before obtaining the hematology values at screening will be excluded.
   2. Hepatic: Total bilirubin ≤ 1.5 times the upper limit of normal (× ULN) (≤ 3 x ULN in the case of Gilbert's disease); Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN (in the case of liver metastases ≤ 5 × ULN); Alkaline phosphatase (ALP) ≤ 2.5 × ULN (≤ 5 × ULN inthe case of liver and/or bone metastases).
   3. Renal: Serum creatinine < 1.5 × ULN or creatinine clearance ≥ 30 mL/min based on Cockcroft-Gault glomerular filtration rate estimation.
   4. Coagulation: International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless on medication known to alter INR and/or aPTT.
   5. Nutritional status: Serum Albumin ≥ 2.8 g/dL.
9. Bisphosphonates or denosumab dosage must have been stable for at least 4 weeks before Day 1 for patients receiving these therapies.
10. Patients must agree to use a condom when is engaged in sexual activity with a pregnant woman during the treatment period and for at least 90 days after last dose of enzalutamide or at least 120 days after last dose of talazoparib (PF-06944076), whichever occurs later. Patients must also agree to use an additional highly effective form of contraception or two effective contraceptive methods, when is engaged in sexual intercourse with a woman of childbearing potential during the treatment period and for at least 90 days after last dose of enzalutamide or at least 120 days after last dose of talazoparib (PF-06944076), whichever occurs later.
11. Must agree to refrain to donate sperm during the treatment period and for at least 90 days after last dose of enzalutamide or at least 120 days after last dose of talazoparib (PF-06944076), whichever occurs later.
12. PSA ≥ 4 ng/mL at diagnosis or before starting ADT therapy.

Exclusion Criteria:

1. Prior treatment with enzalutamide, apalutamide, darolutamide or abiraterone acetate.
2. History of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills.
3. Known hypersensitivity to recombinant proteins, or any excipient contained in the drug formulation for talazoparib (PF-06944076) and enzalutamide.
4. Prior systemic therapy for metastatic prostate cancer (mPCa). Note: Initiation of androgen deprivation therapy (ADT) within 4 weeks prior to study entry would be allowed (with or without first-generation antiandrogens), providing a tumor biopsy sample was taken prior to initiation of ADT is made available for biomarker studies and upon approval by the sponsor. If patient was started on first-generation antiandrogens, these would be discontinued on prior to randomization.

   Note: Patients relapsing after having received an ADT-based regimen in neoadjuvant or adjuvant setting will be suitable for the study if metastatic progression occured while on non-castrate testosterone levels or at least 12 months after discontinuation of ADT.
5. Treatment with approved or investigational cancer therapy within 28 days (or 5 half-lives of the drug- whichever is longer) prior to initiation of study treatment.
6. Known or suspected brain metastases or active leptomeningeal disease.
7. Symptomatic or impending spinal cord compression or cauda equina syndrome.
8. Subject has a history of seizure or any condition that may predispose to seizure (i.e. prior significant brain trauma, brain vascular malformations, ...), or subjects that have had unexplained loss of consciousness or transient ischemic attacks within 1 year prior to scheduled Day 1 of treatment.
9. Therapeutic radiation therapy within 14 days (seven days for limited-field palliative radiotherapy) prior to study enrolment, or patients who have not recovered from radiotherapy-related toxicities to grade ≤ 1 according to National Cancer Insitute ́s Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v.)5.0.
10. Major surgery (defined as requiring general anesthesia) or significant traumatic injury within 14 days of start of study drugs, or patients who have not recovered from the side effects of any major surgery.
11. History of another malignancy within three years of study enrollment with the exception of carcinoma in situ, non-melanoma skin carcinoma, or American Joint Committee on Cancer stage 0 or stage 1 cancer that has a remote probability of recurrence in the opinion of the investigator and the Sponsor's Medical Monitor is required, or any concurrent malignancy for which the patient is receiving therapy.
12. Active uncontrolled infection at the time of enrollment.
13. Congenital long QT syndrome or Electrocardiogram (ECG) at screening with QT interval corrected using Fridericia's formula (QTcF) > 500 milliseconds.
14. Patients with clinically significant cardiovascular disease including but not limited to any of the following:

    1. Stroke, transient ischemic attack, unstable angina pectoris, or documented myocardial infarction within 12 months prior to study entry.
    2. Symptomatic pericarditis or clinically significant pericardial effusion or myocarditis.
    3. Documented congestive heart failure (New York Heart Association functional classification III- IV).
    4. Uncontrolled, persistent hypertension defined as systolic blood pressure > 170 mmHg or diastolic blood pressure > 100 mmHg.
15. Patients have any of the following cardiac conduction abnormalities:

    1. Ventricular arrhythmias except for benign premature ventricular contractions.
    2. Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication.
    3. Conduction abnormality requiring a pacemaker.
    4. Other cardiac arrhythmia not controlled with medication.
16. Patients have any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment contraindicate patient participation in the clinical study.
17. Treatment with estrogens, cyprotoerone acetate or glucocorticoids (at a dose greater than the equivalent to 10 mg/day of prednisone) in the 4 weeks prior to scheduled Day 1 of treatment.
18. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or patients who are employees of the trial sponsor, including their family members, directly involved in the conduct of the study.
19. Concurrent participation in other clinical trial, except other translational studies or observational studies (defined as those with no therapeutic intervention).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Prostate specific antigen complete response (PSA-CR) | Baseline up to 12 months
  The primary efficacy endpoint for the study is the PSA-CR. The PSA-CR is defined as the percentage of patients with PSA < 0.2 ng/mL divided by the number of patients in the analysis set.

SECONDARY OUTCOMES:
Efficacy determined by Prostate specific antigen complete response (PSA-CR) | Baseline up to 7 months
  PSA-CR is defined as the number of patients with PSA <0.2 ng/mL from randomization to Cycle 7 Day 1 therapy divided by the number of patients in the analysis set.
Efficacy determined by PSA response | Baseline up to 7 and 12 months
  PSA response is defined as the number of patients with PSA <0.4 ng/mL from randomization to 7- or 12-months therapy divided by the number of patients in the analysis set
Efficacy determined by Time to Clinical Progression (TCP) | Baseline up to 12 months
  TCP is defined as the time from randomization to clinical progression, based on progression in bone as per 2+2 rule, progression per RECIST criteria v1.1. or clinical deterioration due to cancer per investigator's opinion.
Efficacy determined by Prostate-Specific Antigen progression of disease (PSA-PD) | Baseline up to 12 months
  PSA-PD in accordance with PCWG3 criteria, is defined as the time from randomization to PSA progression.
Efficacy determined by Prostate-Specific Antigen progression-free survival (PSA-PFS) | Baseline up to 12 months
  PSA-PFS in accordance with based on Prostate Cancer Working Group 3 (PCWG3) criteria (PSA ≥ 25% and ≥ 2 ng/mL from nadir confirmed by a second value obtained 3 or more weeks later).
Efficacy determined by Radiological progression-free survival (rPFS) | Baseline up to 12 months
  PFS is defined as the time from randomization to radiological progression based on progression in bone as per 2+2 rule or progression per RECIST criteria v1.1.
Efficacy determined by Time to development of castration resistant (TTCR) prostate cancer | Baseline up to 12 months
  TTCR prostate cancer is defined as the time from randomization to PSA progression in accordance with PCWG3 criteria or clinical progression, whichever occurred first.
Efficacy determined by Overall survival (OS) | Baseline up to 12 months
  OS is defined as the time from randomizatiom date to date of death due to any cause or the last date the patient was known to be alive.
Incidence of adverse events (AEs) | Up to 53 months after study start
  Incidence of prespecified AEs as per National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v.5.0, change from baseline in targeted vital signs, and change from baseline in targeted clinical laboratory test results.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Mateo, Principal Investigator — VHIO
Locations (8):
- Spain (8):
  - Institut Català d'Oncologia Badalona, Badalona
  - Hospital Clínic i Provicial de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Universitario Miguel Sevet, Zaragoza